CLINICAL TRIAL: NCT03869177
Title: Implementation of Guidelines on Family Involvement for Persons With Psychotic Disorders in Community Mental Health Centres. A Cluster Randomised Controlled Trial.
Brief Title: Implementation of Family Involvement for Persons With Psychotic Disorders.
Acronym: IFIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo Metropolitan University (Other); University Hospital, Akershus (Other); Helse Fonna (Other); Diakonhjemmet Hospital (Other); Vestre Viken Hospital Trust (Other); Oslo University Hospital (Other); Sykehuset i Vestfold HF (Other); Sykehuset Telemark (Other Government); The Research Council of Norway (Other); Helse Sor-Ost (Other Government)
Responsible Party: Principal Investigator, Reidar Pedersen, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NFR 262863
Record Dates: First submitted 2019-02-28; First posted 2019-03-11 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Psychotic Disorders
Keywords: Family psychoeducation; Schizophrenia; Implementation science; Mental health care services; Clinical ethics; Family involvement; Family intervention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomised controlled trial. Fourteen clusters will be stratified into three strata according to their estimated number of patients with psychotic disorders currently in treatment. The clusters within each stratum will then be randomised to either intervention or control arms with an allocation ratio of 1:1.The seven outpatient units in the intervention arm receives a comprehensive implementation support program, whereas the outpatient clinics in the control arm receives no implementation support.
  A similar number of patients and relatives will be recruited from both arms, preferably in dyadic pairs, for the quantitative patient- and relative sub study. Employees from the clusters in the intervention arm will be recruited to answer a questionnaire, as part of the implementation study. Patients, relatives and employees will be recruited from the clusters in the intervention arm to take part in qualitative interviews.
Masking Description: Patients and relatives will not be informed about their outpatient clinic's allocation status. However, they may deduce this from the kind of treatment they receive. It's impossible to blind the care providers and for practical reasons we won't be able to blind the investigators or the outcomes assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Other): Clusters (psychiatric outpatient clinics) in the intervention arm receives a comprehensive implementation support program during the trial period.
  Interventions: Other: Implementation support program
- Control arm (No Intervention): Clusters (psychiatric outpatient clinics) in the control arm receives no implementation support during the trial period.

INTERVENTIONS:
Other: Implementation support program — The IFIP intervention consists of the following elements:
  I. Clinical interventions 1.1 A basic level of family involvement and support 1.2 Family psychoeducation in single-family groups
  II. Implementation interventions 2.1 Training and guidance of health care personnel 2.2 A family coordinator 2.3 Other implementation measures
  Arms: Intervention arm

SUMMARY:
This study will develop and evaluate a complex intervention to implement guidelines on family involvement for patients with psychotic disorders (F20-29 in International Classification of Diseases ICD-10) in community mental health centres, by using a cluster randomised design. Fifteen Norwegian outpatient units participate in the study, and each of them constitutes a single cluster, except for two collaborating clinics who are considered one cluster.

Of the fourteen clusters, half will receive implementation support and training immediately, whereas the other half will receive it one and a half year later. The study will assess both service level outcomes, by measuring fidelity scores, and selected outcomes for patients and relatives, by collecting questionnaires and data from central health registers and patient records. In addition, qualitative interviews will be performed with patients, relatives and health care personnel. The study will also include a cost-effectiveness analysis and a political economy analysis.

DETAILED DESCRIPTION:
Background:

Family involvement during severe mental illness, such as psychotic disorders, is both important and challenging. Evidence suggest that family interventions for persons with psychotic disorders are associated with positive outcomes for both relatives and patients, and economic analyses of such interventions consistently report net saving. There are also important moral imperatives to involve those providing unpaid and informal care. Yet research has shown that relatives of patients with severe mental illness experience little involvement, and that the implementation of family interventions is patchy. The Norwegian national guidelines on family involvement in the public health- and care services and the national guidelines on psychotic disorders, both give recommendations on family involvement. However, there is little knowledge about how to achieve their implementation, and whether a high degree of implementation will be associated with improvements in selected outcomes for patients and relatives.

Setting:

Fifteen outpatient units from community mental health centres in the South-Eastern Norway Regional Health Authority.

Research questions:

1. What is the current level of implementation of the selected recommendations in the national guidelines on family involvement for persons with psychotic disorders in participating clinical units?
2. What are important barriers to and facilitators for implementing the national guidelines among the stakeholders at the clinical, organisational, and policy level?
3. What are important moral dilemmas and conflicting interests related to family involvement, and how can these be resolved?
4. Is implementation of the selected recommendations increased by a comprehensive implementation support program, compared with no such support?
5. Is a higher level of implementation of the selected recommendations associated with improvements in selected outcomes for patients and relatives?
6. Is implementation of family involvement during primary psychotic disorders a cost-effective intervention?

Hypotheses:

1. The current implementation of the selected recommendations in the national guidelines on family involvement for persons with psychotic disorders is low.
2. There are important barriers to and facilitators for implementing the national guidelines among the stakeholders, at the clinical, organisational and policy level.
3. There are important moral dilemmas and conflicting interests, and these can be dealt with through systematic triadic approaches and ethics reflection.
4. A comprehensive implementation program for the selected recommendations is associated with a significantly higher implementation of family involvement for persons with psychotic disorders, compared to no such specific program.
5. Higher implementation of the selected recommendations is associated with improved outcomes for patients and relatives.
6. Outcomes for relatives, patients and the public health- and welfare services justify the costs of implementing family involvement for persons with psychotic disorders.

ELIGIBILITY:
Eligibility criteria apply to participants in both quantitative and qualitative sub-studies, except that participation in family psychoeducation as described below is NOT an exclusion criterion in the qualitative sub-study.

Inclusion criteria for patients:

* To have an established psychotic disorder (F20-29 in ICD-10) or a tentative diagnosis of psychotic disorder, certain enough to begin treatment. This need not be the patient's primary diagnosis.
* To be 18 years or older at the time of inclusion.

Exclusion criteria for patients:

* To be sentenced to psychiatric treatment.
* Not being competent to consent to participation in research.
* Having completed more than five joint sessions of family psychoeducation in single-family groups (patient and relative together) or more than ten joint sessions (multiple families together) in multiple-family groups, or a similarly structured family intervention.
* Not having any relatives or next of kin.

Inclusion criteria for relatives:

* Being a relative of a patient with a diagnosis as described above.
* To be 18 years or older at the time of inclusion.

Exclusion criteria for relatives:

• Having completed more than five joint sessions (patient and relative together) of family psychoeducation in single-family groups or more than ten joint sessions (multiple families together) in multiple-family groups, or a similarly structured family intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Implementation study: Fidelity to the intervention model - Family psychoeducation 1 | Baseline, 6, 12 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in score on fidelity scale for performance and content of family psychoeducation. Rated from 1 (low) to 5 (high).
Implementation study: Fidelity to the intervention model - Family psychoeducation 2 | Baseline, 6, 12 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in score on fidelity scale for penetration rate and general organisation of family psychoeducation. Rated from 1 (low) to 5 (high).
Implementation study: Fidelity to the intervention model - Family involvement and support 1 | Baseline, 6, 12 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in total fidelity measured by the fidelity scale for family involvement and support. Rated from 1 (low) to 5 (high).
Implementation study: Fidelity to the intervention model - Family involvement and support 2 | Baseline, 6, 12 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in penetration rate, measured by the fidelity scale for family involvement and support. Rated from 1 (low) to 5 (high).
Implementation study: Fidelity to the intervention model - Family involvement and support 3 | Baseline, 6, 12 and 18 months in the intervention arm. Baseline and 18 months in the control arm.
  Change in content, structure and implementation, measured by the scale for family involvement and support. Rated from 1 (low) to 5 (high).

SECONDARY OUTCOMES:
Patient quantitative sub-study: Patient experiences of their own mental health and functioning. | 0, 6 and 12 months.
  The Behavior and Symptom Identification scale - (BASIS-24) with 24 questions on mental health, functioning and substance use, on a scale 1-5. Completed by patients.
Patient quantitative sub-study and economic sub-study: Quality of life | 0, 6 and 12 months.
  The Recovering Quality of Life - (ReQoL-10) questionnaire with 10 mental health items, and one physical health item on a scale 1-5. Completed by patients.
Patient quantitative sub-study: General satisfaction. | 0, 6 and 12 months.
  The Manchester Short Assesment of Quality of Life - (MANSA) questionnaire - first question only, on a scale 1-7. Completed by patients.
Patient quantitative sub-study: Experienced burden of mental health problems. | 0, 6 and 12 months.
  A single question - Produced for this study on a scale 1-7. Completed by patients.
Patient quantitative sub-study: Perceived warmth and criticism from relative. | 0, 6 and 12 months.
  Hooley 1989 - 5 items rated 1-10. Completed by patients.
Patient quantitative sub-study: Experienced shared decision making. | 0, 6 and 12 months.
  The CollaboRATE questionnaire (3 items rated 0-9), plus two additional items. Completed by patients.
Patient quantitative sub-study: Adherence with medication | 0, 6 and 12 months for patients and relatives. 0 and 12 months for clinicians.
  A single question answered by patient, relative and clinician.
Patient quantitative sub-Study: Clinician assessment of patient mental health and functioning | 0 and 12 months.
  Health of the Nation Outcome Scale - (HoNOS) scale rated by clinicians on 12 items rated 0-4 (no problem - very serious problem).
Patient quantitative sub-study: Clinician assessment of patient global functioning | 0 and 12 months.
  Global Assessment of Functioning Scale - (GAF), split version for symptoms and functioning
Patient quantitative sub-study and economic sub-study: Change in number of hospital admissions. | Measured from 18 months before inclusion to 18 months after inclusion.
  Retrieved from the Norwegian patient registry.
Patient quantitative sub-study and economic sub-study: Change in number of days spent admitted to hospital. | Measured from 18 months before inclusion to 18 months after inclusion.
  Retrieved from the Norwegian patient registry.
Relative quantitative sub-study and economic sub-study: Caregiver quality of life 1 | 0, 6 and 12 months.
  The Care Related Quality of Life - (CarerQoL) questionnaire - Seven questions on a three-point scale. Completed by relatives.
Relative quantitative sub-study and economic sub-study: Caregiver quality of life 2 | 0, 6 and 12 months.
  The Care Related Quality of Life - (CarerQoL) questionnaire - One visual analogue scale (VAS)-question on an 11-point scale, which is also part of the same measure. Completed by relatives.
Relative quantitative sub-study: Experience of caregiving | 0, 6 and 12 months.
  The Experience of Caregiving inventory - (ECI) questionnaire - 66 items on a five-point scale covering various aspects of being a caregiver. Completed by relatives.
Relative quantitative sub-study: Expressed emotion | 0, 6 and 12 months.
  The Family questionnaire - (FQ) - 20 items on a four-point scale, measuring criticism and emotional over-involvement. Completed by relatives.
Relative quantitative sub-study: Experienced involvement and shared decision making | 0, 6 and 12 months.
  An adapted version of the CollaboRATE questionnaire (3 items rated 0-9), plus two additional items completed by relatives.
Relative quantitative sub-study: Experienced support | 0, 6 and 12 months.
  Carer Well-being and Support questionnaire (CWS) v2 short part B - 18 items rated on a four-point scale. Completed by relatives.
Patients' and relatives' quantitative sub-studies and economic sub-study: Use of public health services and resources. | Measured from 18 months before inclusion to 18 months after inclusion.
  Patients' and relatives' use of public health services and resources: Number of appointments with health services, investigations, treatments and medical prescriptions, translated into costs. Retrieved from national registries.
Patients' and relatives' quantitative sub-studies and economic sub-study: Work participation | Measured from 18 months before inclusion to 18 months after inclusion.
  Patients' and relatives' work participation measured in percentage of a regular full time position. Retrieved from national registries.
Economic sub-study: Increased costs related to implementing and practicing family involvement | Measured before baseline and then throughout the implementation period (0-18 months).
  Increased costs related to implementing and practicing family involvement in the clinical units in the intervention arm. Compared to normal costs before baseline.

OTHER OUTCOMES:
Patient quantitative sub-study: Alcohol abuse | 0 months - baseline screening only
  The Alcohol Use Disorders Identification Test - (AUDIT) - 10 items on a five-point scale. Completed by patients.
Patient quantitative sub-study: Drug abuse | 0 months - baseline screening only
  The Drug Use Disorders Identification Test - (DUDIT) - 11 items on a three to five-point scale. Completed by patients.
Patient quantitative sub-study and implementation study: Exposure to family psychoeducation. | Baseline screening, then 6 and 12 months
  Participation in family psychoeducation measured in number and type of sessions. Reported by both patient and clinician.
Relative quantitative sub-study and implementation study: Exposure to psychoeducation. | Baseline screening, then 6 and 12 months
  Participation in family psychoeducation measured in number and type of sessions. Reported by relative.
Relative quantitative sub-study and implementation study: Exposure to family involvement. | Baseline screening, then 6 and 12 months
  Use of different services to involve and support relatives: Family therapy, group support meetings, meetings with the patients' health care personnel, therapy, education on mental health and illness.
Implementation study: Clinician readiness for change | 0, 6 and 12 months, approximately.
  Implementation Process Assessment Tool - (IPAT) a questionnaire (27 items rated 1-6) regarding experience of implementation of a specified practice. Completed by clinicians

CONTACTS AND LOCATIONS:
Overall Officials: Reidar Pedersen, PhD, Principal Investigator — Professor and head of department, Centre for medical ethics,University of Oslo
Locations (15):
- Norway (15):
  - Asker DPS - Vestre Viken HF, Asker
  - Drammen DPS - Vestre Viken HF, Drammen
  - Ringerike DPS - Vestre Viken HF, Hønefoss
  - Kongsberg DPS - Vestre Viken HF, Kongsberg
  - DPS poliklinikk Vestmar/stathelle - Sykehuset Telemark, Kragerø
  - Vestfold DPS - Sykehuset i Vestfold HF, Larvik
  - Nedre Romerike DPS - Akershus Universitetssykehus HF, Lillestrøm
  - Groruddalen DPS - Akershus Universitetssykehus HF, Oslo
  - Søndre Oslo DPS - Oslo Universitetssykehus HF, Oslo
  - Voksenpsykiatrisk avdeling Vinderen - Diakonhjemmet Sykehus, Oslo
  - DPS poliklinikk Porsgrunn - Sykehuset Telemark, Porsgrunn
  - Bærum DPS -Vestre Viken HF, Sandvika
  - DPS poliklinikk Seljord - Sykehuset Telemark, Seljord
  - DPS poliklinikk Skien - Sykehuset Telemark, Skien
  - Vestfold DPS - Sykehuset i Vestfold HF, Tønsberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eisen SV, Normand SL, Belanger AJ, Spiro A 3rd, Esch D. The Revised Behavior and Symptom Identification Scale (BASIS-R): reliability and validity. Med Care. 2004 Dec;42(12):1230-41. doi: 10.1097/00005650-200412000-00010. PMID 15550803
- [Background] Keetharuth AD, Brazier J, Connell J, Bjorner JB, Carlton J, Taylor Buck E, Ricketts T, McKendrick K, Browne J, Croudace T, Barkham M. Recovering Quality of Life (ReQoL): a new generic self-reported outcome measure for use with people experiencing mental health difficulties. Br J Psychiatry. 2018 Jan;212(1):42-49. doi: 10.1192/bjp.2017.10. PMID 29433611
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Background] Szmukler GI, Burgess P, Herrman H, Benson A, Colusa S, Bloch S. Caring for relatives with serious mental illness: the development of the Experience of Caregiving Inventory. Soc Psychiatry Psychiatr Epidemiol. 1996 Jun;31(3-4):137-48. doi: 10.1007/BF00785760. PMID 8766459
- [Background] Brouwer WB, van Exel NJ, van Gorp B, Redekop WK. The CarerQol instrument: a new instrument to measure care-related quality of life of informal caregivers for use in economic evaluations. Qual Life Res. 2006 Aug;15(6):1005-21. doi: 10.1007/s11136-005-5994-6. PMID 16900281
- [Background] Wiedemann G, Rayki O, Feinstein E, Hahlweg K. The Family Questionnaire: development and validation of a new self-report scale for assessing expressed emotion. Psychiatry Res. 2002 Apr 15;109(3):265-79. doi: 10.1016/s0165-1781(02)00023-9. PMID 11959363
- [Background] Quirk, A., Smith, S., Hamilton, S., Lamping, D., Lelliot, P., Stahl, D., Pinfold, V & Andiappan, M. (2012). Development of the carer well-being and support (CWS) questionnaire. Mental Health Review Journal 17:128-38.doi:10.1108/13619321211287184
- [Background] Wing JK, Beevor AS, Curtis RH, Park SB, Hadden S, Burns A. Health of the Nation Outcome Scales (HoNOS). Research and development. Br J Psychiatry. 1998 Jan;172:11-8. doi: 10.1192/bjp.172.1.11. PMID 9534825
- [Background] Berman AH, Bergman H, Palmstierna T, Schlyter F. Evaluation of the Drug Use Disorders Identification Test (DUDIT) in criminal justice and detoxification settings and in a Swedish population sample. Eur Addict Res. 2005;11(1):22-31. doi: 10.1159/000081413. PMID 15608468
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Karterud S, Pedersen G, Løvdal H, Friis S. S-GAF: Global Funsjonsskåring - Splittet Versjon [Global Assessment of Functioning - Split version]. Bakgrunn og skåringsveiledning. Klinikk for psykiatri, Ullevål sykehus, Oslo, 1998.
- [Background] Hooley JM, Teasdale JD. Predictors of relapse in unipolar depressives: expressed emotion, marital distress, and perceived criticism. J Abnorm Psychol. 1989 Aug;98(3):229-35. doi: 10.1037//0021-843x.98.3.229. PMID 2768657
- [Background] Pharoah F, Mari J, Rathbone J, Wong W. Family intervention for schizophrenia. Cochrane Database Syst Rev. 2010 Dec 8;(12):CD000088. doi: 10.1002/14651858.CD000088.pub2. PMID 21154340
- [Background] Yesufu-Udechuku A, Harrison B, Mayo-Wilson E, Young N, Woodhams P, Shiers D, Kuipers E, Kendall T. Interventions to improve the experience of caring for people with severe mental illness: systematic review and meta-analysis. Br J Psychiatry. 2015 Apr;206(4):268-74. doi: 10.1192/bjp.bp.114.147561. PMID 25833867
- [Background] Helsedirektoratet. (2013). Utredning, behandling og oppfølging av personer med psykoselidelser. Retrieved March 22, 2018, from https://helsedirektoratet.no/Lists/Publikasjoner/Attachments/326/Nasjonal-faglig-retningslinje-for-utredning-behandling-og-oppfolging-av-personer-med-psykoselidelser-IS-1957.pdf.
- [Background] Helsedirektoratet. (2017). Veileder om pårørende i helse- og omsorgstjenesten. Retrieved March 22, 2018, from https://helsedirektoratet.no/Retningslinjer/Pårørendeveileder.pdf
- [Background] McHugo GJ, Drake RE, Whitley R, Bond GR, Campbell K, Rapp CA, Goldman HH, Lutz WJ, Finnerty MT. Fidelity outcomes in the National Implementing Evidence-Based Practices Project. Psychiatr Serv. 2007 Oct;58(10):1279-84. doi: 10.1176/ps.2007.58.10.1279. PMID 17914003
- [Background] Vermeulen, B., Lauwers, H., Spruytte, N., Van Audenhove, C., Magro, C., Saunders, J. & Jones, K. (2015). Experiences of family caregivers for persons with severe mental illness: an international exploration. Leuven: LUCAS KU Leuven/EUFAMI.
- [Background] Torrey WC, Drake RE, Dixon L, Burns BJ, Flynn L, Rush AJ, Clark RE, Klatzker D. Implementing evidence-based practices for persons with severe mental illnesses. Psychiatr Serv. 2001 Jan;52(1):45-50. doi: 10.1176/appi.ps.52.1.45. PMID 11141527
- [Background] Campbell MK, Piaggio G, Elbourne DR, Altman DG; CONSORT Group. Consort 2010 statement: extension to cluster randomised trials. BMJ. 2012 Sep 4;345:e5661. doi: 10.1136/bmj.e5661. No abstract available. PMID 22951546
- [Derived] Norheim I, Pedersen R, Selle ML, Rossberg JI, Hestmark L, Heiervang KS, Ruud T, Asholt VM, Hansson KM, Moller P, Fosse R, Kjus SHH, Romoren M. Effectiveness of implementing family involvement on patient outcomes in individuals with psychotic disorders: a pragmatic cluster randomised controlled trial. BMC Psychiatry. 2025 Dec 4;25(1):1142. doi: 10.1186/s12888-025-07501-z. PMID 41345598
- [Derived] Norheim I, Pedersen R, Selle ML, Rossberg JI, Hestmark L, Heiervang KS, Ruud T, Asholt VM, Hansson KM, Moller P, Fosse R, Romoren M. Implementation of guidelines on Family Involvement for persons with Psychotic disorders: a pragmatic cluster randomized trial. Effect on relatives' outcomes and family interventions received. Front Psychiatry. 2024 May 24;15:1381007. doi: 10.3389/fpsyt.2024.1381007. eCollection 2024. PMID 38855639
- [Derived] Hestmark L, Romoren M, Heiervang KS, Hansson KM, Ruud T, Saltyte Benth J, Norheim I, Weimand B, Pedersen R. Implementation of Guidelines on Family Involvement for Persons with Psychotic Disorders (IFIP): A Cluster Randomised Controlled Trial. Adm Policy Ment Health. 2023 May;50(3):520-533. doi: 10.1007/s10488-023-01255-0. Epub 2023 Feb 16. PMID 36797515
- [Derived] Hansson KM, Romoren M, Weimand B, Heiervang KS, Hestmark L, Landeweer EGM, Pedersen R. The duty of confidentiality during family involvement: ethical challenges and possible solutions in the treatment of persons with psychotic disorders. BMC Psychiatry. 2022 Dec 20;22(1):812. doi: 10.1186/s12888-022-04461-6. PMID 36539741
- [Derived] Hansson KM, Romoren M, Pedersen R, Weimand B, Hestmark L, Norheim I, Ruud T, Hymer IS, Heiervang KS. Barriers and facilitators when implementing family involvement for persons with psychotic disorders in community mental health centres - a nested qualitative study. BMC Health Serv Res. 2022 Sep 12;22(1):1153. doi: 10.1186/s12913-022-08489-y. PMID 36096844
- [Derived] Hestmark L, Heiervang KS, Pedersen R, Hansson KM, Ruud T, Romoren M. Family involvement practices for persons with psychotic disorders in community mental health centres - a cross-sectional fidelity-based study. BMC Psychiatry. 2021 Jun 2;21(1):285. doi: 10.1186/s12888-021-03300-4. PMID 34078306
- [Derived] Hestmark L, Romoren M, Heiervang KS, Weimand B, Ruud T, Norvoll R, Hansson KM, Norheim I, Aas E, Landeweer EGM, Pedersen R. Implementation of guidelines on family involvement for persons with psychotic disorders in community mental health centres (IFIP): protocol for a cluster randomised controlled trial. BMC Health Serv Res. 2020 Oct 9;20(1):934. doi: 10.1186/s12913-020-05792-4. PMID 33036605